CLINICAL TRIAL: NCT02604069
Title: Postoperative Monitoring of Tissue Perfusion in Microvascular Free Flaps Using Continuous Interstitial Glucose Monitoring Device: A Pilot Study
Brief Title: Detection of Flap Ischemia Using Interstitial Glucose Monitor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Thoma, Achilleas (Individual); Jiayi Hu (Unknown); Matthew McRae (Unknown)
Responsible Party: Principal Investigator, Ronen Avram, Associate Professor, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CGM-2015-10
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Free Tissue Flaps
Keywords: Breast reconstruction; Breast cancer; Microsurgery; Continuous flap monitor
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Continuous Glucose Monitor (Experimental): Application of CGM for 6 days following free flap reconstruction in conjunction with clinical monitoring
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor

SUMMARY:
A simple device that objectively assesses flap perfusion - either as a stand-alone tool or an adjunct to the current monitoring method - would be a tremendous improvement in detection of early postoperative flap ischemia and, in turn, increase flap salvage and survival. In this study, the investigators aim to examine the accuracy and reliability of measuring interstitial glucose levels using Continuous Glucose Monitoring (CGM) technology as an objective method of detecting postoperative flap tissue ischemia in patients undergoing free flap-based reconstructive surgery.

DETAILED DESCRIPTION:
Background:

Breast reconstruction involving microvascular free tissue transfer is a major, labour-intensive operation that provides numerous benefits for patients' psychosocial function and well-being.

Flap failure, though rare, is a devastating complication and leads to serious morbidities. It can occur in the first 24-72 hours after the operation. However, if ischemia is detected earlier, the chances for operative salvage are better. Unfortunately, the current monitoring process remains mostly subjective.

A simple device that objectively assesses flap perfusion - either as a stand-alone tool or an adjunct to the current monitoring method - would be a tremendous improvement in detection of early postoperative flap ischemia and, in turn, increase flap salvage and survival.

Purpose:

The overall objective of this clinical pilot study is to examine the accuracy and reliability of measuring interstitial glucose levels using Continuous Glucose Monitoring (CGM) technology as an objective method of detecting postoperative flap tissue ischemia in patients undergoing free flap-based reconstructive surgery.

Methods:

In this pilot cohort study, the investigators aim to prospectively include 30 free flaps in total from 10-20 patients undergoing DIEP-based breast reconstruction by one surgeon at Juravinski Hospital. Patients will be recruited at the pre-operative consultation. The transcutaneous sensor of the CGM device will be inserted into the subcutaneous layer of the flap upon completion of surgery, while an additional sensor will be placed on the patient's thigh as control. These devices are blinded and will start recording the flap's interstitial glucose levels. The patient will be admitted and the flap will be assessed clinically as per protocol. On-call residents will be given a data collection sheet to document the exact time they were alerted about a flap, the clinical finding, and the subsequent decision made. Once an endpoint has been reached for a flap, the CGM sensor will be removed and its data extracted.

Data Analysis:

The timing of occurrence of low interstitial glucose levels and rapid glucose level decline will be analyzed with the timing of clinical concerns raised about the flap. The systemic glucose level will be used as a control for the flap glucose level. The investigators aim to analyze the temporal correlation between interstitial glucose measurements and clinical findings of the flap's vascular status (eg. vessel occlusion, ischemia). Statistical analysis will be done with assistance by a biostatistician.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing unilateral or bilateral breast reconstruction with free flap including DIEP flaps at Hamilton Health Sciences, starting from the date of ethics approval.

Exclusion Criteria:

* Patients with diabetes (on oral antiglycemic medications or insulin-dependent)
* Patients who are on immunosuppressive medication
* Patients undergoing breast reconstruction involving expanders or implants
* Patients with active infections

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Temporal correlation between interstitial glucose measurements and flap ischemia | within 6 days after surgery

SECONDARY OUTCOMES:
Incidence of minor side effects related to device | within 6 days after surgery
Incidence of major adverse effects related to the device | within 6 days after surgery
Incidences of technical issues related to the device | within 6 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Avram, MD, Principal Investigator — Associate Professor, Plastic Surgery
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada